CLINICAL TRIAL: NCT02858024
Title: A Two-Cohort, Open-Label, Randomised, Three-Period Crossover Trial In Healthy HIV-Negative Women To Assess The Effect Of Menses And Tampon Use On The Pharmacokinetics Of Dapivirine, Delivered By Dapivirine Vaginal Ring-004, Containing 25 Mg Of Dapivirine
Brief Title: A Trial In Healthy HIV-Negative Women To Assess The Effect Of Menses And Tampon Use On The Pharmacokinetics Of Dapivirine, Delivered By Dapivirine Vaginal Ring-004, Containing 25 Mg Of Dapivirine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IPM 035
Record Dates: First submitted 2016-07-19; First posted 2016-08-08 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: HIV

ARMS (2):
- Cohort I (Active Comparator): In Cohort I, eligible participants will be randomly assigned to one of two treatment sequences (ABE or BAE). During two consecutive 28-day treatment periods (treatment periods 1 and 2), separated by a washout period of 28 days, the participants will receive each of the following treatments according to their assigned treatment sequence
  Interventions: Drug: Dapivirine Vaginal Ring-004 and no tampons; Drug: Dapivirine Vaginal Ring-004 with tampons; Drug: Dapivirine Vaginal Ring-004 with no menses
- Cohort II (Active Comparator): In Cohort II, eligible participants will be randomly assigned to one of two treatment sequences (CDE or DCE). During two consecutive 28-day treatment periods (treatment periods 1 and 2), separated by a washout period of 28 days, the participants will receive each of the following treatments according to their assigned treatment sequence
  Interventions: Drug: Dapivirine Vaginal Ring-004 with no menses; Drug: Dapivirine Vaginal Ring-004 and same ring inserted after menses; Drug: Dapivirine Vaginal Ring-004 and new ring inserted after menses

INTERVENTIONS:
Drug: Dapivirine Vaginal Ring-004 and no tampons — Dapivirine Vaginal Ring-004 for 28 days, with menses, no tampon use (Treatment A),
  Other Names: Treatment A
  Arms: Cohort I
Drug: Dapivirine Vaginal Ring-004 with tampons — followed by Dapivirine Vaginal Ring-004 for 28 days, with menses, with tampon use (Treatment B)
  Other Names: Treatment B
  Arms: Cohort I
Drug: Dapivirine Vaginal Ring-004 with no menses — Dapivirine Vaginal Ring-004 for 28 days, with no menses occurring (Treatment E; treatment period 3).
  Other Names: Treatment E
Drug: Dapivirine Vaginal Ring-004 and same ring inserted after menses — Dapivirine Vaginal Ring-004 used continuously until the start of menses, at which time the ring will be removed, and the same ring re-inserted five days later (estimated completion of menses) (Treatment C)
  Other Names: Treatment C
  Arms: Cohort II
Drug: Dapivirine Vaginal Ring-004 and new ring inserted after menses — Dapivirine Vaginal Ring-004 used continuously until the start of menses, at which time the ring will be removed, and a new ring inserted five days later (estimated completion of menses) (Treatment D)
  Other Names: Treatment D
  Arms: Cohort II

SUMMARY:
A Two-Cohort, Open-Label, Randomised, Three-Period Crossover Trial In Healthy HIV-Negative Women To Assess The Effect Of Menses And Tampon Use On The Pharmacokinetics Of Dapivirine, Delivered By Dapivirine Vaginal Ring-004, Containing 25 Mg Of Dapivirine

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible to enroll in the trial:

1. Women 18 and ≤ 40 years of age who can give written informed consent;
2. Available for all visits and consent to follow all procedures scheduled for the trial;
3. Healthy, based on medical history, vital signs, physical examination, urinalysis (dipstick and microscopy [if indicated]), laboratory evaluations for genital infections (bacterial vaginosis, gonorrhoea, chlamydia, and trichomonas), and laboratory evaluations for haematology and biochemistry;
4. HIV-negative as determined by an HIV test at screening;
5. On a stable oral contraceptive regimen for at least three months prior to screening;
6. Upon pelvic examination at the time of enrollment, the cervix and vagina appear normal as determined by the Investigator/Physician;
7. Asymptomatic for genital infections at the time of enrollment (if a woman is diagnosed with any treatable STI, either clinically or by laboratory test at the time of screening, she must have completed treatment before the date of enrollment);
8. Willing to refrain from the use of topical vaginal medications, vaginal products or objects, including female condoms, cotton wool, rags, diaphragms, cervical caps (or any other vaginal barrier method), douches, lubricants, vibrators/dildos, and drying agents for seven days prior to enrollment and for the duration of the trial;
9. Willing to refrain from tampon use during menses for the entire duration of the trial, other than when assigned to Treatment B (Cohort I);
10. Documentation of no abnormality on cervical cytology, including grossly bloody smear, within 90 days prior to screening;
11. Willing to refrain from participation in any other research trial for the duration of this trial;
12. Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures, e.g. by home visit or telephone, or via family or close neighbor contacts (confidentiality to be maintained);
13. Willing to agree to abstain from all the following for a total of 2 days (48 hours) prior to each trial visit; Penile-vaginal intercourse Oral contact with her genitalia
14. Hepatitis B and C negative at the time of enrollment.

Exclusion Criteria:

Participants who meet any of the following criteria are NOT eligible to enrol in the trial:

1. Currently pregnant or had their last pregnancy outcome within three months prior to screening;
2. Currently breast-feeding;
3. Currently or within two months of participation in any other clinical research trial involving investigational or marketed products prior to screening;
4. Untreated symptomatic urogenital infections, e.g. urinary tract or other STIs, or other gynaecological conditions such as vaginal itching, pain, or discharge, within two weeks prior to enrollment;
5. Have a Grade 2 or higher pelvic examination finding, according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events; Addendum 1 Female Genital Grading Table for Use in Microbicide Studies;
6. History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, urethral obstruction, incontinence or urge incontinence;
7. Current vulvar or vaginal symptoms/abnormalities that could influence the trial results;
8. Cervical cytology at screening that requires cryotherapy, biopsy, treatment (other than for infection), or further evaluation;
9. Symptomatic genital herpes simplex virus (HSV) infection or a history of genital herpetic infection;
10. Any Grade 2, 3 or 4 haematology, biochemistry or urinalysis laboratory abnormality at baseline (screening) according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events; Addendum 1 Female Genital Grading Table for Use in Microbicide Studies;
11. Unexplained, abnormal bleeding per vagina during or following vaginal intercourse, or gynaecologic surgery within 90 days prior to enrollment;
12. Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex or silicone;
13. Any serious acute, chronic or progressive disease (e.g. any known history of neoplasm, cancer, diabetes, epilepsy, cardiac disease, autoimmune disease, HIV, AIDS, or blood dyscrasias), or signs of cardiac disease, renal failure, or severe malnutrition;
14. Have undergone a hysterectomy and/or bilateral oophorectomy and/or presented with amenorrhea within 90 days prior to enrollment;
15. Any condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2016-04-16 (Actual); Study Completion 2016-04-16 (Actual)

PRIMARY OUTCOMES:
Dapivirine concentrations in vaginal fluid and in plasma, measured at specified time points before, during, and after menses, when no tampons are used, during a 28-day ring use period. | 28 days
  To determine the effect of menses on the local and systemic pharmacokinetics (PK) of dapivirine, delivered by the Dapivirine Vaginal Ring-004, in healthy, HIV-negative women
Dapivirine concentrations in vaginal fluid and in plasma, measured at specified time points before, during, and after menses, when tampons are used, during a 28-day ring use period. | 28 days
  To determine the effect of tampon use during menses on the local and systemic PK of dapivirine, delivered by the Dapivirine Vaginal Ring-004, in healthy, HIV-negative women.

SECONDARY OUTCOMES:
Dapivirine concentrations in vaginal fluid and in plasma, measured at specified time points before, during, and after menses when the ring is removed at the onset of menses, and re-inserted after completion of menses for the remainder of a 28-day period. | 28 days
  To assess the impact on the local and systemic PK of dapivirine, delivered by the Dapivirine Vaginal Ring-004 when the ring is removed at the start of menses, and re-inserted after completion of menses.
Dapivirine concentrations in vaginal fluid and in plasma, measured at specified time points before, during, and after menses when the ring is removed at the onset of menses, and a new ring inserted after completion of menses | 28 days
  To assess the impact on the local and systemic PK of dapivirine, delivered by the Dapivirine Vaginal Ring-004 when the ring is removed at the start of menses, and a new ring inserted after completion of menses.
The residual amounts of dapivirine in used vaginal rings, removed at the onset of menses, where applicable, or on Day 28. | 28 days
  To assess residual levels of dapivirine in used rings.
Safety will be assessed through the reporting of AEs, including SAEs, laboratory safety assessments (haematology, biochemistry, and urinalysis), physical and gynaecological examinations, and vaginal flora and pH assessments during the trial. | 28 days
  To assess the safety of the Dapivirine Vaginal Ring-004 in healthy, HIV-negative women.